CLINICAL TRIAL: NCT04106713
Title: Understanding the Person, Exploring Change Across Psychotherapies
Acronym: Xchange
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Mental Health, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/01184
Record Dates: First submitted 2019-09-16; First posted 2019-09-27 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Depression; Anxiety Disorders
Keywords: Psychotherapy; Cognitive behavioural therapy; Group psychotherapy; Internet-based psychotherapy
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Individual Therapy (Experimental): The individual therapy program will differ in orientation according to therapist and session notes will be coded according to the Comparative Psychotherapy Process Scale. Therapy sessions take place approximately once every fortnight, with 8 sessions in total, according to the agreed-upon schedule.
  Interventions: Behavioral: Individual Psychotherapy
- Internet-delivered Cognitive Behavioural Therapy (iCBT) (Experimental): The iCBT program (clinician follow-up with the therapist and 4 online modules) will be administered for 8 weeks. The four modules: "1) psychoeducation about emotions, including a functional nature of emotions; 2) alteration of antecedent cognitive misappraisals; 3) prevention of emotional avoidance; and 4) modification of emotion-driven [behaviours] (EDBs)", are adapted from The Unified Protocol (UP) for transdiagnostic treatment of emotional disorders. UP is a CBT consisting of four overarching themes- "increasing emotional awareness, facilitating flexibility in appraisals, identifying and preventing [behavioural] and emotional awareness, and situational and interoceptive exposure to emotion cues".
  Interventions: Behavioral: Internet-delivered Cognitive Behavioural Therapy (iCBT)
- Group CBT (Experimental): The group CBT program (for e.g. PsychUp) will be conducted over 8 weeks, with weekly 2-hour sessions. Each group consists of 4-8 patients and are facilitated by two practicing clinical psychologists and one clinical psychologist in training. Sessions are structured such that each session, except the first, begins with a brief review of previous session material and a collaborative review of homework. This is followed by introduction of new material and completion of any in-session exercises, with sessions concluding with homework assignment. Specific treatment content is similarly adapted from UP. Session 1 begins by covering psychoeducation on the CBT model of pathological depression and anxiety and the role of avoidance in maintenance of symptoms. Sessions 2 to 7 covers goal-setting, cognitive reappraisal and development of adaptive emotional coping strategies through situational emotion-focused exposures. Session 8 ends with a discussion on relapse prevention.
  Interventions: Behavioral: Group Cognitive Behavioural Therapy (group CBT)
- Delayed Waitlist (No Intervention): Participants in the Waitlist group will be recruited from those referred for psychotherapy and who are not assigned to either group or iCBT and not planned for psychotherapy at IMH for 8 weeks or more from the point of consent.
- Treatment as Usual (TAU) (No Intervention): Participants in the Treatment as Usual (TAU) group are individuals who are not assigned to psychotherapy at IMH. They will be recruited from outpatient services and emergency services at IMH.

INTERVENTIONS:
Behavioral: Individual Psychotherapy — The individual therapy program will differ in orientation according to therapist and session notes will be coded according to the Comparative Psychotherapy Process Scale. Therapy sessions take place approximately once every fortnight, with 8 sessions in total, according to the agreed-upon schedule.
  Arms: Individual Therapy
Behavioral: Internet-delivered Cognitive Behavioural Therapy (iCBT) — The iCBT program (clinician follow-up with the therapist and 4 online modules) will be administered for 8 weeks. The four modules: "1) psychoeducation about emotions, including a functional nature of emotions; 2) alteration of antecedent cognitive misappraisals; 3) prevention of emotional avoidance; and 4) modification of emotion-driven [behaviours] (EDBs)", are adapted from The Unified Protocol (UP) for transdiagnostic treatment of emotional disorders. UP is a CBT consisting of four overarching themes- "increasing emotional awareness, facilitating flexibility in appraisals, identifying and preventing [behavioural] and emotional awareness, and situational and interoceptive exposure to emotion cues".
  Arms: Internet-delivered Cognitive Behavioural Therapy (iCBT)
Behavioral: Group Cognitive Behavioural Therapy (group CBT) — The group CBT program (for e.g. PsychUp) will be conducted over 8 weeks, with weekly 2-hour sessions. Each group consists of 4-8 patients and are facilitated by two practicing clinical psychologists and one clinical psychologist in training. Sessions are structured such that each session, except the first, begins with a brief review of previous session material and a collaborative review of homework. This is followed by introduction of new material and completion of any in-session exercises, with sessions concluding with homework assignment. Specific treatment content is similarly adapted from UP. Session 1 begins by covering psychoeducation on the CBT model of pathological depression and anxiety and the role of avoidance in maintenance of symptoms. Sessions 2 to 7 covers goal-setting, cognitive reappraisal and development of adaptive emotional coping strategies through situational emotion-focused exposures. Session 8 ends with a discussion on relapse prevention.
  Arms: Group CBT

SUMMARY:
Identifying predictors and understanding mechanisms of change will inform referral to psychotherapy, triage and right-siting by helping clinicians to understand how their patients are likely to benefit from clinical interventions. This study will be the first of its kind conducted in an Asian hospital setting to identify the predictors of response to individual, group and internet-delivered CBT for the treatment of depressed and anxious patients in the Institute of Mental Health (IMH), Singapore. With increasing challenges with hospital workload, there is an increasing emphasis on group and online interventions. Understanding of the factors that may predict outcome from these therapies can improve right-siting by identifying who will get better without therapy or who may not benefit from a given form of therapy and guide personalisation of care. An important biological predictor of outcome is likely to be genetic risk as it has been demonstrated that patients with greater melancholia and a family history may not be sufficiently treated with brief courses of therapy. Identifying psychological factors underlying psychological distress and determining the extent to which these factors are addressed by these interventions will help to improve and individualise existing psychotherapy and motivate new psychotherapeutic interventions.

DETAILED DESCRIPTION:
All IMH outpatients who have been referred for psychotherapy will be invited to take part in this research. Participants will be recruited from triage, outpatient clinics, emergency services and referrals from therapists. In specific, participants under the iCBT and group CBT (for e.g. PsychUp) treatment arms will be recruited from the Psychology Department from triage and those under individual therapy will be recruited from the Psychotherapy Department.

After indicating interest to participate in the study, potential patients will be contacted to explain the purpose of the study and its procedures, obtain informed consent to take part in the study as well as brief them on how to log on and access and complete questionnaires.

Participants will be placed into the study arms (i.e. iCBT, group CBT or individual therapy) based on the intervention program each has been allocated to. Some participants will also form a Delayed Waitlist group. Other participants will form the Treatment as Usual (TAU) group. Participants in the Waitlist group will be recruited from those referred for psychotherapy and who are not assigned to either group or iCBT and not planned for psychotherapy at IMH for 8 weeks or more from the point of consent. Participants in the Treatment as Usual (TAU) group are individuals who are not assigned to psychotherapy at IMH. They will be recruited from outpatient services and emergency services at IMH.

The Waitlist and Treatment as Usual Groups will serve as the control groups.

For all groups, psychiatric and medical history, pharmacological and other non-psychological interventions will first be obtained at baseline in order to control for other treatment effects. Such medical records would be accessed via c-Doc; data will be obtained from information management and the IMH diagnostics. SAP data at IMH, including demographic data, postal code, diagnosis, race, clinician names (but not limited to), will be collected for this study.

For the psychotherapy arms (iCBT, group CBT, and individual therapy), assessments will be conducted from baseline across the course of participants' psychotherapy interventions as well as into follow-up. A baseline battery will be completed before the start of therapy. The baseline battery includes vulnerability measures, around half of which will serve as the independent variables and the other half will be used to assess outcome, during their first visit (i.e. triage). This series of baseline measures will take approximately 50 min to complete. For iCBT, group CBT and individual therapy, there will be study visits after each session of therapy, whereby participants will be asked to complete a series of additional measures. The series of weekly measures will take approximately 15 min to complete. Any measures that the therapists use regularly when sending out the measures will be left out and the therapist can request for the outcomes to be either emailed or uploaded on C-doc for their reference. After the last session, participants would complete a post-intervention battery besides the post-session measures. The series of post-intervention measures, to be completed above the weekly measures on the last therapy session, will take approximately 45 min to complete.

Mechanisms of change: Process-outcome in Individual Therapy In 30 clients undergoing frequent individual therapy (ideally once a fortnight or more), in addition to the quantitative measurement of outcome, consent will be taken to allow audio with or without video recording of their sessions. Their therapist will also provide consent for recording of sessions. Sessions will be recorded by their therapist. Sessions will be subsequently transcribed and coded with scales to assess alliance-building, interventions, and emotional work. Initial coding will use the comparative psychotherapy process scale, the facilitative interpersonal scale, and the emotional arousal scale according to a coding manual by trained raters.

For every 3 months for two years (if consented to), participants may complete the follow-up measures. For iCBT and group CBT, therapy sessions would take place weekly for 8 weeks. For individual therapy, therapy sessions take place approximately once every fortnight, with 8 sessions in total, according to the agreed-upon schedule.

Buccal swabs will be obtained from consenting participants at baseline and post-therapy to conduct genome-wide association scanning to construct polygenic risk scores for prediction of response to therapy and assess epigenetics as a vulnerability factor pre-post therapy.

Timeline and list of measures for waitlist and group TAU (refer to appendix): For waitlist/TAU, assessments will be completed at Week 0, Week 4, Week 8 and for follow-ups (see attached Gantt chart).

Participants in the waitlist/ TAU groups will not undergo buccal swabs.

Participants in the waitlist arm would be individuals who have been referred for psychotherapy but would not be undergoing therapy for at least 8 weeks from the point of recruitment into this study, and hence will serve as the control group. It is highly likely that a considerable proportion of participants in the waitlist group would eventually undergo therapy within the period of study follow up (up to 2 years). In this case, the data collected from such participants from before they begin therapy would first be retained, and such participants would also subsequently be recruited into the psychotherapy arm of the study, where they would complete all procedures of the study.

In the event that TAU participants are referred for psychotherapy over the duration of the study, the data collected from such participants from before they begin therapy would first be retained, and also subsequently recruit them into the psychotherapy arm of the study.

Baseline and post-intervention measures will be completed online.

For post-session/ follow-up measures online, Pragmatic Tracker, an official online platform used by the Institute of Mental Health for administering scales to therapy patients, will be utilized. Any measures that the therapists use regularly will be left out when sending out the measures and the therapist can request for the outcomes to be either emailed or uploaded on Cdoc for their reference.

For all groups, psychiatric and medical history, pharmacological and other non-psychological interventions will first be verified during follow-up in order to control for other treatment effects. Such medical records would be accessed via c-Doc. Data will be obtained from information management and the IMH diagnostics.

Like the therapists, the triage psychologists will also be given a background information form during triage review that probes their experience as a triage officer and general client expectations (Therapist/Triage Officer Background Information Form). It is hypothesized that such evaluations by the triage psychologists may affect treatment outcome. For TAU and Waitlist, the patient's clinician will assist in completing the GAF.

Incidental findings are not anticipated for any patients from this study. Only DNA will be extracted after the collection of the buccal swabs, which would not reveal any incidental findings of potential health and reproductive importance. However, the possibility that a genetic test will be developed in the future that can use the collected data and predict the development of a disease in later life with certainty, and which becomes apparent from the study's analyses, cannot be excluded. This is considered to be unlikely as the study only looks at common genetic variants in this study. The study informs participants of the potential to uncover incidental findings in future research in the ICF, and provide for re-identification of participants in such cases.

There will not be any incidental findings for the therapists as there will not be any biological/clinical tests that the therapists themselves will complete that may reveal potential health or reproductive importance.

Hard copies or soft copies of scales may be administered at all time points or may be administered over the phone, depending on the preference on the participants and licensing permissions. Scales will be made available for completion online wherever possible, except for scales such the Anxiety Sensitivity Index (only allowed to be administered on paper) and EQ5D-L5 (on phone/ paper). Online modes of administration include Pragmatic Tracker, REDCAP and QuestionPro. QuestionPro and REDCAP are research platforms also used by IMH/SICS and have the function of scheduling surveys at several time points.

ELIGIBILITY:
Inclusion Criteria:

1. For patients:

   1. 18-99 years old;
   2. have current or past symptoms of anxiety and/or depression;
   3. able to communicate and read in English;
   4. able to provide informed consent.
   5. Waitlist arm:

      - Referred for psychotherapy but given a waiting time of 8 weeks or more to the first visit or not assigned to therapy at IMH.
   6. Treatment as usual:

      - Not assigned to any psychotherapeutic interventions.
   7. iCBT: - Referred for iCBT;

      - Identified as a 'P2' patient/appropriate for iCBT by triage.
   8. Group therapy:

      - Referred for group therapy;

      - Identified as a 'P2' patient/appropriate for group therapy by triage.
   9. Individual psychotherapy:

      * Referred for individual therapy;
      * Patient and therapist committed to frequent therapy (ideally fortnightly).
2. For therapists:

   1. Therapists who will see OR have been assigned to clients in the waitlist arm, iCBT, group therapy (e.g. PsychUp), and individual psychotherapy group.

Exclusion Criteria:

1. For patients:

1. current active suicidal intention or plan;
2. cognitively-impaired/are unable to consent/lack capacity to consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) score | Immediately before each therapy session for 8 sessions (i.e. 8 weeks for iCBT and group therapy, or approximately 16 weeks for individual therapy), and at follow-up every 3 months up to 2 years.
  Depression scale. Total scores range from 0 to 27, with higher scores representing more severe depression.
Change in Generalized Anxiety Disorder-7 (GAD-7) questionnaire score | Immediately before each therapy session for 8 sessions (i.e. 8 weeks for iCBT and group therapy, or approximately 16 weeks for individual therapy), and at follow-up every 3 months up to 2 years.
  Anxiety scale. Total scores range from 0 to 21, with higher scores representing more severe anxiety.
Change in Outcome Rating Scale (ORS) score | Immediately before each therapy session for 8 sessions (i.e. 8 weeks for iCBT and group therapy, or approximately 16 weeks for individual therapy).
  Measure assessing general well-being. Total scores range from 0 to 40, with higher scores representing better general well-being.
Change in Work and Social Adjustment Scale (WSAS) score | At baseline, at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy), and at follow-up every 3 months up to 2 years.
  The WSAS is a self-report scale of functional impairment attributable to an identified problem. Total scores range from 0 to 40, with higher scores representing greater functional impairment.

SECONDARY OUTCOMES:
Change in Self-Referential Encoding Task (SRET) performance | At baseline, at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy), and at follow-up every 3 months up to 2 years.
  The SRET is a computerized task which involves a self-descriptive judgment phase where participants respond to trait adjectives presented as describing or not describing them, followed by a later recall phase where they attempt to remember the words presented. Only the self-descriptive judgment phase will be included in this study. Words from an SRET validated in predicting depressive relapse, the Revised Interpersonal Adjective Scales: Big Five Version (IASR-B5), as well as words based on the life events used in the LEC, will be incorporated into the SRET as the trait adjectives used in the self-descriptive judgment phase. The self-descriptive judgment phase of the SRET, as a measure of negative implicit self-referential cognition, is associated strongly with depression.
Change in Implicit Association Task (IAT) performance | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The IAT is a computerized task which can be used to measure subconscious associations between mental representations of different concepts. For this study, it is designed specifically to assess attitudes towards therapy.
Change in Partner Go/No Go Association Task (P-GNAT) performance | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The P-GNAT is a computerized task which is an implicit measure assessing personal evaluations of another individual. For this study, it is designed specifically to assess attitudes towards the therapist.
Change in Go/No Go Association Task (GNAT) performance | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The GNAT is a computerized task to assess inhibitory control and processing speed.
Change in Letter-number Sequencing Task performance | At baseline, and at post-intervention (immediately after the final and final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  Computerized task to assess working memory capabilities.
Change in Word Fluency Task performance | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  Computerized task to assess verbal functioning.
Change in Cognitive Style Questionnaire-Very Short Form (CSQ-VSF) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The CSQ-VSF measures negative cognitive styles. Scores range from 7 to 35 on both the Globality subscale and Stability subscale, 10 to 50 on the Negative consequences subscale, and 3 to 15 on the Self-woth implications subscale, with higher scores representing more negative cognitive style. Subscale scores are summed to obtain the total score.
Change in Leiden Index of Depression Sensitivity-Revised Revised(LEIDS-RR) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The LEIDS-RR measures cognitive reactivity to sadness across the domains of acceptance/coping (ACC), avoidant coping (AVC), perfectionism/control (CTR), aggression (AGG), and hopelessness/suicidality (HOP). Scores range from 0 to 24 on the ACC and AGG subscales, 0 to 32 on the AVC subscale, and 0 to 20 on the CTR and HOP subscales, with higher scores representing greater cognitive reactivity. Subscale scores are summed to obtain the total score.
Change in Reconstructed Depressive Experiences Questionnaire (RecDEQ) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The RecDEQ measures and differentiates between the anaclitic (dependent) and introjective (self-critical) types of depression, with introjective depression associated with perfectionism. Scores range from 10 to 70 on the anaclitic depression subscale and 9 to 63 on the introjective depression subscale, with higher scores representing more severe depression.
Change in Dysfunctional Attitudes Scale (DAS-24) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The DAS-24 measures maladaptive patterns of thinking. Scores range from 8 to 56 each on the Achievement, Self-control, and Dependence subscales, with higher scores representing greater maladaptive patterns of thinking.
Change in Anxiety Sensitivity Index (ASI) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The ASI measures tendency to fear the physical and cognitive symptoms associated with anxiety. Total scores range from 0 to 64 with higher scores representing greater fear of symptoms associated with anxiety.
Change in Person's Relating to Others Questionnaire (PROQ3) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  PROQ3 measures people's interpersonal difficulties in the form of negative and maladaptive relating to others. It comprises of 8 scales, upper neutral (UN); upper close (UC); neutral close (NC); lower close (LC); lower neutral (LN); lower distant (LD); neutral distant (ND); and upper distant (UD), based upon the eight octants of a theoretical structure called the interpersonal octagon. Scores on each of these subscales range from 0 to 15, with higher scores representing greater interpersonal difficulties. Subscale scores can be summed to obtain the total score.
Change in Difficulties in Emotion Regulation Scale Short Form (DERS-SF) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The DERS-SF measures problems with emotion regulation across six domains of non-acceptance of emotional responses (Non-acceptance subscale), difficulties engaging in goal-directed behavior (Goals subscale), impulse control difficulties (Impulse subscale), lack of emotional awareness (Awareness subscale), limited access to emotion regulation strategies (Strategies subscale), and lack of emotional clarity (Clarity subscale). Scores range from 3 to 15 on each of the subscales, with higher scores representing greater difficulty with emotional regulation. Subscale scores can be summed to obtain the total score.
Change in Inventory for Depressive Symptomatology (IDS) scores | At baseline (IDS-30), at post-intervention (QIDS-16) (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy), and at follow-up every 3 months up to 2 years (QIDS-16).
  The IDS-30 measures severity of depressive symptoms. Melancholic depression can be identified via an algorithm involving a selected 9 items of the IDS-30.
  The Quick Inventory of Depressive Symptomatology-16 (QIDS-16) is a shorter version derived from the IDS-30. QIDS-16 total scores are highly correlated with, and can be converted to, IDS-30 total scores.
Change in Generalized Anxiety Disorder-7 (GAD-7) questionnaire score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  Anxiety scale. Total scores range from 0 to 21, with higher scores representing more severe anxiety. An additional open-ended question will query what stimuli usually results in the anxiety.
Change in Patient Health Questionnaire-Panic Disorder (PHQ-PD) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  Measures frequency and severity of panic attacks. Total scores range from 0 to 15, with higher scores representing greater frequency or severity of panic attacks.
Change in Positive Mental Health Instrument (PMH) scores | At baseline (PMH-Short), at post-intervention (PMH-Short) (immediately after final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy) and at follow-up every 3 months up to 2 years (PMH-Rapid)
  The PMH measures mental health and well-being. The PMH-Short and PMH-Rapid are shorter versions derived from the PMH. Total scores can be converted to a range from 1 to 6, with higher scores representing more positive mental health.
Change in EuroQol 5-dimension 5-level (EQ-5D-5L) Descriptive System scores | At baseline, and at follow-up every 3 months up to 2 years.
  The EQ-5D-5L Descriptive System measures five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has scores ranging from 1 to 5, with higher scores representing poorer quality of life.
Change in EuroQol 5-dimension 5-level (EQ-5D-5L) Visual Analogue Scale scores | At baseline, and at follow-up every 3 months up to 2 years.
  The EQ-5D-5L Visual Analogue Scale measures perception of one's current health on a scale of 0 to 100, with higher scores representing better health.
Change in modified Clinical Global Impression (self-report) scores | At baseline, at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy), and at follow-up every 3 months up to 2 years.
  The modified CGI measures severity of illness (on a scale of 1 to 7, higher scores representing greater severity), global improvement (on a scale of 1 to 7, 1= Very much improved, 4 = no change, 7 = Very much worse), state of recovery (from 0% to 100% recovered) and the efficacy of treatment (on a scale of 1 to 16, with higher scores representing lower efficacy).
Change in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) scores | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The Q-LES-Q-SF measures quality of life. Total scores range from 16 to 80, with higher scores representing better quality of life.
Change in Frequency of Actions and Thoughts Scale (FATS) score | Immediately after each therapy session (i.e. over 8 weeks for iCBT and group therapy, or over approximately 16 weeks for individual therapy), at post-intervention (immediately after final session), and at follow-up every 3 months up to 2 years.
  The FATS measures patients' application of adaptive skills that have been taught during therapy. Total scores range from 0 to 48, with higher scores representing greater frequency of application of adaptive skills.
Change in Clinical Outcomes in Routine Evaluation-10 (CORE-10) score | Immediately after therapy session for 8 sessions (i.e. over 8 weeks for iCBT and group therapy, and approximately 16 weeks for individual therapy)
  The CORE-10 is a brief clinical outcome measure with total scores ranging from 0 to 40. Higher scores represent better clinical outcomes.
Change in Working Alliance Inventory-Short Revised (WAI-SR) | Immediately after each therapy session for 8 sessions (i.e. 8 weeks for iCBT and group therapy; approximately 16 weeks for individual therapy).
  The WAI-SR measures patient's perceptions of alliance in psychotherapy. Total scores range from 12 to 60, with higher scores representing better working alliance.
Feedback Questionnaire | Immediately after each therapy session for 8 sessions (i.e. 8 weeks for iCBT and group therapy; approximately 16 weeks for individual therapy).
  A short open-ended questionnaire regarding patients' feedback on therapy. This questionnaire will consist of two Likert scale ratings (from 1-5) assessing patients' perception of how useful and how relevant the week's session was to their problems, followed by three open-ended questions for patients to elaborate on their feedback and specify particular aspects of the session (i.e., "What did you find to be the most helpful component of therapy this week?", "What did you find to be less or not helpful this week?", "What do you think can be improved this week?"). This questionnaire is aimed at obtaining consistent session-by-session feedback from patients that will further facilitate the focus groups.
Session Rating Scale (SRS) | Immediately after each therapy session for 8 sessions (i.e. 8 weeks for iCBT and group therapy; approximately 16 weeks for individual therapy).
  The SRS is a four-item visual analogue scale designed to assess key dimensions of effective therapeutic relationships. Total scores range from 0 to 40, with higher scores representing more effective therapeutics relationships.
Default rates | During intervention (8 sessions, i.e. over 8 weeks for iCBT and group therapy, or over approximately 16 weeks for individual therapy).
  The proportion of patients who default or terminate early from therapy.
Change in Psychodynamic Functioning Scale (PFS) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The PFS is a therapist-completed measure that assesses patients in 6 dimensions: 1. Quality of Family Relations, 2. Quality of friendships, 3. Romantic/sexual relationships, 4. Tolerance for affects, 5. Insight, 6. Problem solving and adaptive capacity. Each dimension is rated on a scale of 0 to 100, with higher scores representing better outcomes.
Change in Global Assessment of Functioning (GAF) score | At baseline, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The GAF is a therapist-completed measure that assesses the social, occupational and psychological functioning of a client. Total scores range from 0 to 100, with higher scores representing better functioning.
Change in Working Alliance Inventory-Short Revised-Clinician (WAI-SR-C) score | Immediately after the first therapy session, and at post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The WAI-SR-C measures therapist's perceptions of alliance in psychotherapy. Total scores range from 10 to 50, with higher scores representing better working alliance.

OTHER OUTCOMES:
Personality Inventory for DSM-5-Brief Form (PID-5-BF) | At baseline.
  The PID-5-BF measures pathological personality traits in 5 dimensions: negative affect, detachment, antagonism, disinhibition, and psychoticism. Each subscale score ranges from 4 to 20, with higher scores representing a greater degree of each trait.
Eysenck Personality Questionnaire-Revised Short Form Neuroticism Scale (EPQ-R-S-N) | At baseline.
  The EPQ-R-S-N measures neuroticism as a personality trait. Total scores range from 0 to 12, with higher scores representing higher levels of neuroticism.
Life Experiences Checklist (LEC) | At baseline, and at follow-up every 3 months up to 2 years.
  Assesses the number and types of stressful life events experienced, as well as the degree of stress experienced in each.
Childhood Trauma Questionnaire (CTQ) | At baseline.
  The CTQ measures traumatic events in childhood across the types of death of a loved one, parental conflict, victim of physical violence, illness or injury, sexual abuse, and others. Responses for each type of trauma are measured on 2 scales: 1. severity of trauma, 2. degree of confiding in others about the traumatic experience. Scores range from 1 to 7 on each scale, with higher scores representing greater severity of trauma or greater degree of confiding respectively.
Experiences in Close Relationships Questionnaire-12 (ECR-12) | At baseline.
  ECR-12 measures people's adult attachment styles across two dimensions: Attachment Avoidance and Attachment Anxiety. Subscale scores range from 6 to 42, with higher scores indicating greater attachment avoidance or attachment anxiety respectively.
Adult Rejection Sensitivity Questionnaire (A-RSQ) | At baseline.
  The A-RSQ measures people's sensitivity to perceived and actual rejection. Average computed scores range from 1 to 6, with a higher score representing greater sensitivity to rejection.
Comparative Psychotherapy Process Scale (CPPS) | At post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  The CPPS measures the activity, process and techniques used by therapists, over 2 dimensions: Psychodynamic-interpersonal (PI) and Cognitive-behavioral (CB). Subscale scores each range from 0 to 60, with higher scores indicating that the therapy session is more characteristic of that particular therapy modality.
Client Task Specific Change Measure Revised (CTSCM-R) | At post-intervention (immediately after the final therapy session i.e. at 8 weeks for iCBT and group therapy, or at approximately 16 weeks for individual therapy).
  A measure of a client's outcomes. Total scores range from 16 to 112, with higher scores representing better outcomes.
Cooper-Norcross Inventory of Preferences (CNIP) | At baseline.
  The CNIP measures patients' initial preferences of psychotherapy on 4 continuums: Therapist Directiveness vs. Client Directiveness, Emotional Intensity vs. Emotional Reserve, Past Orientation vs. Present Orientation, and Warm Support vs. Focused Challenge. Item scores range from -3 to 3, with greater scores representing a preference for the former end of the continuum.
Credibility and Expectancy Questionnaire (CEQ) | At baseline.
  The CEQ measures patients' treatment expectancy and thoughts of rationale credibility regarding psychotherapy. The credibility subscale scores range from 3 to 27, with higher scores representing greater treatment rationale credibility. The expectancy subscale score is derived from a composite score of 3 questions, with higher scores representing greater expectancy.
Client Motivation for Therapy Scale (CMOTS) | At baseline.
  The CMOTS measures patients' motivation for psychotherapy across 6 domains: intrinsic motivation, integrated regulation, identified regulation, introjected regulation, external regulation, and amotivation. Each of these subscales scores range from 4 to 28, with higher scores representing greater motivation.
Readiness for Psychotherapy Index (RPI) | At baseline.
  The RPI measures patients' positive attitude and preparedness for psychotherapy. Total scores range from 20 to 100, with higher scores representing greater readiness for psychotherapy.
Medication Adherence Rating Scale (MARS) | At baseline.
  MARS is a ten-item self-report measure of medication adherence. Total scores range from 0 to 10, with higher scores representing poorer adherence to medication. This scale will be used to control for the nuisance variable of non-psychotherapeutic, medical interventions.
Sociodemographics (self-report) | At baseline.
  A short self-report questionnaire regarding patients' sociodemographics. This questionnaire will consist of items querying their gender, age, socioeconomic status, educational attainment, living arrangement, relationship status, engagement in undesirable habits and physical health.
Psychiatric history (self-report) | At baseline.
  A short self-report questionnaire regarding patients' past psychiatric history. This questionnaire will consist of items querying the number of previous episodes of depression and/or anxiety, the duration of these prior episodes, resultant role impairment, previous engagement in therapy and/or medication and family history of mental illness.
Treatment history/current treatment interventions | At baseline, and at follow-up every 3 months up to 2 years.
  A short questionnaire querying treatment history/ current interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey CY Tan, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Institute of Mental Health, Singapore, Singapore, Singapore